CLINICAL TRIAL: NCT04043338
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Single Ascending Dose Study Investigating the Safety, Tolerability, and Pharmacokinetics of XC130-A10H in Healthy Adult Subjects
Brief Title: Single Ascending Dose Study Investigating the Safety, Tolerability, and PK of XC130-A10H in Healthy Adult Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xoc Pharmaceuticals (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XC130-A10H-CL-101
Record Dates: First submitted 2019-07-24; First posted 2019-08-02 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- XC130-A10H (Experimental): XC130-A10H (single dose)
  Interventions: Drug: XC130-A10H
- Placebo (Placebo Comparator): placebo (single dose)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XC130-A10H — XC130-A10H supplied as a 0.2, 0.4, 0.8, 1.6 or 3.2 mg dose, administered in capsules or tablets
  Arms: XC130-A10H
Drug: Placebo — Placebo supplied as matching capsules or tablets
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group single ascending dose (SAD) study. Up to 5 cohorts of 8 subjects (6 active and 2 placebo) are planned for evaluation. In each cohort, subjects will receive a single oral dose of XC130-A10H or matching placebo on Day 1. Safety, tolerability, and pharmacokinetics will be assessed throughout the study. Dose escalation will not take place until the Principal Investigator, Sponsor, and Medical Monitor have determined that adequate safety and tolerability from the previous cohorts have been demonstrated to permit proceeding to the next cohort.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel group SAD study conducted at one study center. Up to 5 cohorts of 8 subjects (6 active and 2 placebo) are planned for evaluation. In each cohort, subjects will receive a single oral dose of XC130-A10H or matching placebo on Day 1. Dose escalation will not take place until the Principal Investigator, Sponsor, and Medical Monitor have determined that adequate safety and tolerability from the previous cohorts have been demonstrated to permit proceeding to the next cohort.

Safety (i.e., adverse events [AEs], physical examinations, pulse oximetry, vital signs, orthostatic vital signs, 12-lead electrocardiograms (ECGs), clinical laboratory tests, Columbia suicide severity rating scale [C-SSRS], and Mini-Mental State Examination [MMSE]) will be assessed throughout the study. Blood samples will be collected through 48 hours post-dose for the PK assessment of XC130-A10H and the metabolites.

ELIGIBILITY:
Major Inclusion Criteria:

* Healthy, adult, male or female of non-childbearing potential only, 18-75 years of age.
* Body mass index (BMI) ≥ 18 and ≤ 32.0 kg/m2 at screening.
* Medically healthy with no clinically significant findings from medical history, physical examination, laboratory profiles, vital signs or ECGs.
* Understands the study procedures in the informed consent form (ICF), and is willing and able to comply with the protocol.

Major Exclusion Criteria:

* Mental or legal incapacitation or significant emotional problems either present at the time of the screening visit or expected during the conduct of the study.
* History or presence of clinically significant medical, surgical or psychiatric condition or disease.
* History of any illness that, in the opinion of the PI, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
* History of clinically significant hypotension.
* History of orthostatic hypotension in the 12 months prior to screening.
* Clinically significant hypertension at screening.
* History or presence of alcoholism within the 2 years prior to dosing or any history of drug abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2019-08-11 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events | pre-dose through 14 days post-dose
  Adverse Events will be monitored throughout confinement in the clinic and through the 14-day follow-up visit.
Changes from baseline in systolic and diastolic blood pressure | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48 hours
  Blood pressure (systolic and diastolic) will be measured pre-dose and throughout the study at the time points specified and compared to baseline.

SECONDARY OUTCOMES:
Maximum plasma concentration [Cmax] of XC13-A10H | 48 hours
  Blood samples will be collected pre-dose, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 18, 24, and 48 hours post-dose and the maximum observed concentration for XC130-A10H and primary metabolite will be calculated.
Area under the curve [AUC] of XC130-A10H | 48 hours
  Blood samples will be collected pre-dose, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 18, 24, and 48 hours post-dose and the area under the concentration-time curve, from time 0 to the last observed non-zero concentration will be calculated for XC130-A10H and primary metabolite.
Time to reach the maximum plasma concentration [Tmax] of XC130-A10H | 48 hours
  Blood samples will be collected pre-dose, 0.5, 1, 1.5, 2, 3, 4, 8, 12, 18, 24, and 48 hours post-dose and the time to reach the maximum plasma concentration of XC130-A10H and primary metabolite will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Fishman, MD, Study Director — Xoc Consulting Chief Medical Officer
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No